CLINICAL TRIAL: NCT05973253
Title: Evaluation of Efficacy and Safety of Topical 1% Medroxyprogesterone in the Corneal Epithelium Healing After Photorefractive Keratectomy in Feiz Hospital, Isfahan, 2023
Brief Title: Evaluation of Efficacy and Safety of Topical 1% Medroxyprogesterone in the Corneal Epithelium Healing After PRK
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Isfahan Ophthalmology Research Center (Network)
Responsible Party: Principal Investigator, Alireza Peyman, Dr. Alireza Peyman, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.MUI.MED.REC.1402.114
Record Dates: First submitted 2023-07-26; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Photorefractive Keratectomy
Keywords: PRK; MEDROXY PROGESTRONE
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eyes that recieved medroxy progestrone at the end of surgery (Experimental): eyes that received one drop of medroxy progesterone at the end of the photorefractive keratectomy(PRK)
  Interventions: Drug: prepared drop of medroxy progestrone acetat 1%
- eyes did not recieved moderxy progestrone (No Intervention): eyes that did not receive drop medroxy progesterone at the end of photorefractive keratectomy(PRK)

INTERVENTIONS:
Drug: prepared drop of medroxy progestrone acetat 1% — In 37 patients who are candidates for photorefractive keratectomy, at the end of the procedure, in one eye randomly, in addition to the antibiotic drop that is routinely placed at the end of the procedure, a drop of prepared medroxyprogesterone is also placed. Then, a bandage contact lens is placed on the eyes, and the patient receives the routine post-procedure drops that include betamethasone and ciprofloxacin drops for both eyes.
  Other Names: depo provera
  Arms: eyes that recieved medroxy progestrone at the end of surgery

SUMMARY:
In this clinical trial, it is decided that 30 patients who are candidates for photorefractive keratectomy will receive a drop of prepared medroxyprogesterone randomly in one of their eyes, in addition to the routine antibiotic drop that is normally placed at the end of the procedure. Afterward, a bandage contact lens will be applied to both eyes, and the patients will receive routine post-procedure drops, including betamethasone and ciprofloxacin drops for both eyes. On the first, second, third, fourth, and fifth days after the operation, the patients will be examined, and the size of the epithelial defect in both eyes will be assessed using a slit lamp device. Additionally, the patients' pain levels in each eye will be evaluated using a questionnaire."

The main question is: General purpose:

Determining the efficacy and safety of 1% topical medroxyprogesterone in repairing the corneal epithelium after photorefractive keratectomy (PRK)

DETAILED DESCRIPTION:
Patients who have referred for refractive surgery to correct myopia and myopia-stigmatism first undergo complete examinations that are required before the procedure, which includes the following examinations:

1. manifest and cycloplegic refraction
2. UCVA and BCVA
3. Pentacam(topographic imaging)
4. Examining the anterior and posterior segments of the eye with a slit lamp device Placed. Then, on the day of the surgery, in the refractive surgery operating room, the eyes are prepared . Anesthetizing drops of enstocaine are poured into the eyes. After removing the corneal epithelium, laser ablation is performed using the Technolas Teneo 317 device, and then mitomycin C is placed on the cornea based on the amount of ablation and then washed. At the end of the procedure, a contact lens bandage is placed on the eyes, and then a drop of the antibiotic ciprofloxacin is poured into the eyes. At this stage, a 1% medroxyprogesterone drop will be randomly poured into one of the eyes. After discharge, ciprofloxacin and betamethasone drops are routinely prescribed for the patient every 4 hours, and the patient returns for examination on the day after the operation and on the third and fifth days after the operation. (7) In each visit, the size of the corneal epithelial defect is measured by an ophthalmologist with a slit lamp examination as the largest length of the defect and the largest perpendicular length in millimeters. (2) Regarding the patient's pain and discomfort, a questionnaire is used to score the pain intensity by the patient (0: no pain, 1: mild pain, 2: moderate pain, 3: severe pain, 4: unbearable pain). (8) and the checklist includes information: pain intensity, optical size Defect, gender, age, ablation rate, and refractive error will be checked and recorded.

The patient and the examiner do not know about the eye in which medroxyprogesterone drops were used at the end of the procedure.

Medroxyprogesterone drops are made by a pharmacologist under sterile conditions and delivered the day before the operation.

ELIGIBILITY:
Inclusion Criteria:

* 1- Age above 18 years 2- Myopia and myopic astigmatism 3- The stability of the patient's refraction over the past year 4-- Not using contact lenses at least 3 weeks before the operation 5- Absence of history of KCN and any type of corneal ectasia in the patient himself or his first degree family 6- Full satisfaction and knowledge of patients to enter the plan 7- No history of previous eye surgery and eye trauma 8- Absence of active eye diseases, corneal dystrophy, retinal diseases, glaucoma, dry eyes of any degree.

  9- Absence of systemic diseases that can potentially interfere with wound healing, including diabetes, vascular collagen diseases, and pregnancy.

  10- Not taking inhaled or systemic steroids actively or within 3 months before the procedure

Exclusion Criteria:

1. The patient's lack of consent to continue the study
2. Failure to visit the patient for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Determining the efficacy and safety of 1% topical medroxyprogesterone in repairing the corneal epithelium after photorefractive keratectomy (PRK) | 3 months
  Determining the efficacy and safety of 1% topical medroxyprogesterone in repairing the corneal epithelium after photorefractive keratectomy (PRK)

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Peyman, MD, Study Chair — Isfahan ophthalmology research centre
Locations (2):
- Iran (2):
  - Isfahan eyes research centre, Isfahan
  - Isfahan Eye Research Center, Isfahan

IPD SHARING:
Plan to Share IPD: No
Will be shared upon request